CLINICAL TRIAL: NCT06971848
Title: Evaluation of Skin Tests in Biotherapy Allergies
Acronym: ETCABIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC24_0373
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck; Melanoma Neoplasms; Small Cell Bronchial Carcinomas; Bronchial Carcinoma; Pleural Mesothelioma; Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Follicular Lymphoma; Myeloma; AL Amyloidosis; Hepatocarcinoma; Colorectal Cancer; Esophageal Squamous Cell Carcinoma; Heart Cancer; Cholangiocarcinoma; Colorectal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Bronchogenic; Mesothelioma, Malignant; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis; Carcinoma, Hepatocellular; Colorectal Neoplasms; Esophageal Squamous Cell Carcinoma; Heart Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental)
  Interventions: Other: Drug skin tests (investigating hypersensitivity to a biotherapy)

INTERVENTIONS:
Other: Drug skin tests (investigating hypersensitivity to a biotherapy) — allergologic skin tests (prick tests and intradermal tests)

SUMMARY:
Biotherapies are biological (extracted from an organism or living tissue) or biotechnological drugs used in the treatment of multiple conditions, such as autoimmune inflammatory diseases, cancers, and hematologic diseases. In recent years, these biotherapies have notably emerged in the treatment of cancers and hematologic disorders. As such, most patients with cancers or hematologic diseases will likely receive a biotherapy as part of their care pathway.

These biotherapies are associated with various side effects, including hypersensitivity or allergic reactions, which are often poorly characterized in clinical trials. These reactions manifest as symptoms without specific dermatologic or allergologic semiology (such as itching, erythema, shortness of breath, sometimes digestive issues, or discomfort, and in some cases, an anaphylactic reaction).

Unlike other treatments, such as antibiotics and neuromuscular blockers, there are currently no guidelines on the concentrations to use in skin tests for biotherapies. We propose conducting prospective clinical research to scientifically establish the concentrations to be used when investigating hypersensitivity to a biotherapy, in line with best practice recommendations for drug skin testing.

ELIGIBILITY:
Inclusion Criteria :

* Patient treated with one of the biotherapies under study (Atezolizumab 1200 mg, Nivolumab 480 mg, Obinutuzumab 100 mg, Durvalumab 1500 mg, Pembrolizumab 200 mg, Daratumumab 1800 mg, Cemiplimab 3500 mg) and who has received at least two injections of the biotherapy without suspected allergic side effects.
* Subjects covered by or having the rights to medical care assurance
* Written informed consent obtained from subject
* If applicable, treatment with corticosteroids and H1 antihistamines by systemic route (IV or oral) which may be discontinued at least one week before performing the tests (Inhaled corticosteroids are allowed).

Exclusion Criteria:

* Presence of local or diffuse dermatological lesions (e.g., psoriasis, eczema, ...) that could interfere with the interpretation of skin tests.
* Poor understanding of the French language
* Pregnancy, breastfeeding
* Persons in detention by judicial or administrative decision
* Person admitted to a health or social establishment for purposes other than research
* Person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
maximum usable concentration considered non-irritant | Day 1
  For each biotherapy studied, the maximum usable concentration considered non-irritant is defined as the maximum concentration that does not produce a skin reaction in at least 9 out of 10 patients (90% specificity) during skin testing.

SECONDARY OUTCOMES:
possible occurrence of a delayed reaction at 48 hours post-testing | Day 2
  delayed reaction is considered if, at the intradermal injection sites, a skin reaction occurs 48 hours after injection, or if a systemic reaction occurs following biotherapy administration.
possible occurrence of a delayed reaction at one week post-testing | Day 7
  delayed reaction is considered if, at the intradermal injection sites, a skin reaction occurs 1 week after injection

CONTACTS AND LOCATIONS:
Overall Officials: Martine MORISSET, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No